CLINICAL TRIAL: NCT01593735
Title: A Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-2748 in Hepatitis C-Infected Participants
Brief Title: A Multiple Dose Study to Evaluate the Safety and Efficacy of MK-2748 in Hepatitis C-Infected Participants (MK-2748-002 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2748-002; 2011-006296-18 (EudraCT Number)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — MK-2748

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Panel A: GT1, low dose (Experimental): Participants with genotype 1 (GT1) Hepatitis C Virus (HCV) will receive low dose MK-2748 daily for 7 days.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel B: GT1, lower dose (Experimental): Participants with GT1 HCV will receive lower dose MK-2748 daily for 7 days.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel C: GT1, dose based on Panels A+B (Experimental): Participants with GT1 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panels A (low dose) and B (lower dose).
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel G: GT1, dose based on Panels A+B+C (Experimental): Participants with GT1 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panels A (low dose), B (lower dose), and C.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel H: GT1, dose based on Panels A+B+C+G (Experimental): Participants with GT1 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panels A (low dose), B (lower dose), C, and G.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel D: GT3, low dose (Omitted) (Experimental): Participants with genotype 3 (GT3) HCV were to receive low dose MK-2748 daily for 7 days. Panel D was omitted from the study design and participants were not enrolled in this panel.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel E: GT3, high dose (Experimental): Participants with genotype 3 (GT3) HCV will receive high dose MK-2748 daily for 7 days.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel F: GT3, dose based on Panel E (Experimental): Participants with GT3 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panel E (high dose).
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel I: GT3, dose based on Panels E+F (Experimental): Participants with GT3 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panels E (high dose) and F.
  Interventions: Drug: MK-2748; Drug: Placebo
- Panel J: GT3, dose based on Panels E+F+I (Experimental): Participants with GT3 HCV will be dosed with MK-2748 daily for 7 days based on the safety, pharmacokinetic, and/or pharmacodynamic data from Panels E (high dose), F, and I.
  Interventions: Drug: MK-2748; Drug: Placebo

INTERVENTIONS:
Drug: MK-2748 — MK-2748 tablets, orally, once daily for 7 days, dose level dependent on Panel assignment
Drug: Placebo — Placebo tablets, orally, once daily for 7 days

SUMMARY:
This is a multiple dose study of the safety and efficacy of MK-2748 to be done in 2 Parts. Part I will enroll genotype 1 (GT1) hepatitis C virus (HCV)-infected participants and Part II will enroll genotype 3 (GT3) HCV-infected participants. Both Parts may run concurrently or may be staggered.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of chronic HCV infection (GT1 or GT3) for at least 6 months and detectable HCV-RNA in peripheral blood
* Body mass index (BMI) of 18 to 37 kg/m^2
* No clinically significant abnormality on electrocardiogram (ECG)
* Stable health
* Willing to use appropriate contraception throughout the study and for 90 days after last dose of study drug

Exclusion criteria:

* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal (excepting HCV infection), cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic disease (exceptions of adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix, or other malignancies which have been successfully treated ≥10 years prior and unlikely to recur
* Positive Hepatitis B surface antigen
* Documented human immunodeficiency virus (HIV) infection
* Consumption of excessive amounts of alcohol, defined as greater than 2 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces],wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day
* Consumption of excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) or coffee, tea, cola, or other caffeinated beverages per day
* Major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to study enrollment
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Current regular user (including "recreational use") of any illicit drugs or history of drug (including alcohol) abuse within approximately 2 months prior to enrollment
* Evidence or history of chronic hepatitis not caused by HCV including but not limited to non-HCV viral hepatitis, non-alcoholic steatohepatitis (NASH), drug induced hepatitis, autoimmune hepatitis
* Previous treatment with other HCV NS3/4A protease inhibitors
* Previous exposure to interferon-alpha and/or ribavirin within 3 months prior to study enrollment
* Clinical or laboratory evidence of advanced or decompensated liver disease; evidence of bridging fibrosis or higher grade fibrosis (Metavir score ≥3)
* Participation in another investigational study within 4 weeks prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HCV RNA viral load (log 10 copies/mL) in GT1 HCV-infected participants | Predose on Day 1 through Day 56
Change from baseline in HCV RNA viral load (log 10 copies/mL) in GT3 HCV-infected participants | Predose on Day 1 through Day 56
Number of participants experiencing clinical or laboratory adverse events (AEs) | From first dose up to 21 days
Number of participants discontinued from study treatment due to AEs | From Day 1 through Day 7

SECONDARY OUTCOMES:
Area under the plasma concentration curve from Hour 0 to Hour 24 (AUC0-24hr) for MK-2748 | Day 1 and Day 7, predose through 24 hours post-dose
Plasma concentration of MK-2748 (C24) on Day 7 of dosing | 24 hours post-dose on Day 7